CLINICAL TRIAL: NCT00781521
Title: A Pilot, Multicenter, Open Label, Non Comparative Study of the Safety and Efficacy of Floxin Otic Solution in the Treatment of Acute Otitis Media Twice Daily for Seven Days in Children With Tympanostomy Tubes
Brief Title: Safety and Efficacy of Floxin Otic Solution in the Treatment of Acute Otitis Media in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Director Regulatory Affairs, Daiichi Sankyo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8280A-PRT021
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Floxin otic solution twice a day for 7 days
  Interventions: Drug: ofloxacin otic solution 0.3%

INTERVENTIONS:
Drug: ofloxacin otic solution 0.3% — ofloxacin otic solution 0.3% instilled twice a day for seven days

SUMMARY:
This was a pilot study to determine the safety and effectiveness of a twice daily, seven-day dosing regimen in acute, pediatric, otitis media in children with tympanostomy tubes. The currently approved regimen is twice daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 6 months of age to <12 years of age
* weight = or >4.5 kg
* Patent tympanostomy tube(s) in the affected ear(s)
* Purulent or mucopurulent otorrhea of recent onset of presumed bacterial origin

Exclusion Criteria:

* Non-bacterial otic infection
* Known or suspected hypersensitivity to ofloxacin
* Cystic fibrosis
* HIV infection
* Neutropenia
* Receiving immunosuppressive therapy

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2002-11; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Sponsor determined clinical cure of otitis media | 7 days
Sponsor determined microbiological cure of otitis media | 7 days

SECONDARY OUTCOMES:
Investigator determined clinical cure | 7 days
Overall per-subject microbiological outcome | 7 days
Overall per pathogen microbiological outcome | 7 days
sign and symptoms of otitis media | 7 days